CLINICAL TRIAL: NCT03278080
Title: Development of Assessment Method of Driving Ability Using Driving Simulator in Healthy Volunteers #1: Measurement Setup of Assessment Criteria for Driving Ability
Brief Title: Development of Assessment Method for Driving Ability Using Driving Simulator in Healthy Volunteers #1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nagoya University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DS-204-01; JapicCTI-173714 (Other: JapicCTI)
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2017-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- driving test (Other)
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test

INTERVENTIONS:
Other: Road-tracking test — Driving with simulator program for SDLP measurement
Other: Car-following test — Driving with simulator program for DCV measurement
Other: Harsh-braking test — Driving with simulator program for BRT measurement

SUMMARY:
The purpose of this study is to set an optimal measurement time for assessing driving ability in a driving simulator in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and <25.0 kg/m2 at screening inspection
* No visual impairment (enable to correct the vision with eyeglasses or contact lens)
* Receive a prior explanation on the study, able to accept its content, and capable to provide voluntary written consent for participation in this study

Exclusion Criteria:

* History of drug and food allergy
* Routinely drink alcohol before bedtime
* Inappropriate for enrollment in this study was judged by principal investigator or subinvestigator

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) | 60 min.

SECONDARY OUTCOMES:
Distance Coefficient of Variation (DCV) | 25 min.
Brake Reaction Time (BRT) | 15 min.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Fukuoka, Japan